CLINICAL TRIAL: NCT01490788
Title: A Single-Dose, Open-Label, Randomized, Three-Way Crossover Study of the Comparative Bioavailability of TNX-102 2.4 mg and Cyclobenzaprine 5 mg Tablets and of the Effect of Food on the Pharmacokinetics of TNX-102 2.4 mg in Healthy Adults
Brief Title: A Comparative Bioavailability and Pharmacokinetic Study of TNX-102 2.4 mg and Cyclobenzaprine 5 mg Tablets in Healthy Adults.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tonix Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TNX-CY-F101
Record Dates: First submitted 2011-12-07; First posted 2011-12-13 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — cyclobenzaprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): 1 x TNX-102 2.4 mg gelcap under fasting conditions
  Interventions: Drug: Treatment A
- Treatment B (Experimental): 1 x cyclobenzaprine 5 mg immediate release (IR) tablet under fasting conditions
  Interventions: Drug: Treatment B
- Treatment C (Active Comparator): 1 x TNX-102 2.4 mg gelcap under fed conditions
  Interventions: Drug: Treatment C

INTERVENTIONS:
Drug: Treatment A — TNX-102 2.4 mg - 1 gelcap once under fasting conditions.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment A
Drug: Treatment B — Cyclobenzaprine 5 mg, 1 tablet once under fasting conditions
  Other Names: cyclobenzaprine HCl
  Arms: Treatment B
Drug: Treatment C — TNX-102 2.4 mg, 1 gelcap once given under fed conditions.
  Other Names: cyclobenzaprine HCl
  Arms: Treatment C

SUMMARY:
The trial is designed to assess the safety and tolerability of TNX-102 2.4 mg and to compare the bio-availability of TNX-102 2.4 mg and cyclobenzaprine 5 mg tablets under fasting or fed conditions.

DETAILED DESCRIPTION:
Single-center, randomized, open-label, single-dose, three-way-crossover trial is designed to assess the safety and tolerability of TNX-102 2.4 mg (a dose based on the results of a previous Phase 2a, proof-of-concept study - VPI-CY-0001.1) and to compare the rate and extent of absorption of TNX-102 2.4 mg and cyclobenzaprine 5 mg tablets under fasting or fed conditions.

ELIGIBILITY:
Inclusion Criteria: Healthy adults

* Male or female
* Non-smoker
* 18-55 years old
* BMI > 18.5 and < 30.0
* With medically acceptable form of contraception (female only).

Exclusion Criteria:

* Any clinically significant abnormality or vital sign abnormalities
* Any abnormal laboratory test
* History of alcohol or drug abuse or dependence within 1 year and/or positive drug, cotinine, or alcohol tests
* Use of any drug (within 30 days), supplement, or food (within 14 days) known to induce or inhibit hepatic drug metabolism prior to study medication
* Positive pregnancy test, breastfeeding or lactating
* Use of medication other than hormonal contraceptives or topical products, including OTC, natural health products, MAO inhibitors
* Participation in an investigational study within 30 days prior to dosing
* Donation of plasma (within 7 days), or donation or loss of blood of 50-499 mL (within 30 days), or of > 499 mL (within 56 days) prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-11-18; Primary Completion 2011-12-30 (Actual); Study Completion 2011-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Audet, MD, Principal Investigator — PharmaNet
Locations (1):
- PharmaNet, Inc., Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment A First, Then B, Then C: Single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions), Washout (7 days), Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions), Washout (7 days), Single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions)
- Treatment A First, Then C, Then B: Single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions), Washout (7 days), Single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions), Washout (7 days), Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions)
- Treatment B First, Then A, Then C: Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions), Washout (7 days), single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions), Washout (7 days), single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions)
- Treatment B First, Then C, Then A: Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions), Washout (7 days), single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions), Washout (7 days), single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions)
- Treatment C First, Then A, Then B: Single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions), Washout (7 days), single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions), Washout (7 days), Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions)
- Treatment C First, Then B, Then A: Single dose of Treatment C (2.4 mg TNX-102 gelcap under fed conditions), Washout (7 days), Single dose of Treatment B (5 mg cyclobenzaprine IR tablet under fasting conditions), Washout (7 days), single dose of Treatment A (2.4 mg TNX-102 gelcap under fasting conditions)
Period: Overall Study
Arm/Group | Treatment A First, Then B, Then C | Treatment A First, Then C, Then B | Treatment B First, Then A, Then C | Treatment B First, Then C, Then A | Treatment C First, Then A, Then B | Treatment C First, Then B, Then A
Started | 5 | 5 | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5 | 5 | 5
Not Completed | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All subjects that were randomized to receive all three treatments.
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Region of Enrollment [Number; unit: participants]
  Canada | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Concentration (AUC) of Cyclobenzaprine
Description: Blood samples were collected pre-dose, 30 min, 1, 1.5, 2, 2.5, 3, 3.33, 3.67, 4, 4.67, 5, 5.5, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose for each treatment period.
Time Frame: 0 to 96 hours
Measure: Mean (Full Range); unit: pg.hr/mL
Groups:
- Treatment A: All study subject who were administered one TNX-102 2.4 mg gelcap under fasting conditions during the course of the study.
- Treatment B: All study subject who were administered one IR tablet of cyclobenzaprine 5 mg under fasting conditions during the course of the study.
- Treatment C: All study subject who were administered one TNX-102 2.4 mg, gelcap under fed conditions during the course of the study.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 30 | 30 | 30
pg.hr/mL | 47,074.19 [30288.11 to 63860.27] | 94,874.26 [60588.45 to 129160.07] | 50,263.16 [30725.75 to 69800.57]

2. Primary Outcome: Incidences of Adverse Events
Description: Every adverse events occurring during the study period will be reported.
Time Frame: Continuously until the end (day 5) of each study period + 8-10 days after end of last period (total duration: about 1 month)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 30 | 30 | 30
Participants
  Subjects with Treatment-Emergent Adverse Events | 14 | 15 | 10
  Subjects with Serious Adverse Events | 0 | 0 | 0
  Subjects discontinued due to adverse event | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 months
Groups:
- Treatment C: All study subject who were administered one TNX-102 2.4 mg gelcap under fed conditions during the course of the study.
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 14/30 | 15/30 | 10/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=30) | Treatment B (N=30) | Treatment C (N=30)
Palpitations (Cardiac disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 1
Blood Pressure increased (Investigations) | 2 | 1 | 1
Somnolence (Nervous system disorders) | 3 | 11 | 2
Ear Discomfort (Ear and labyrinth disorders) | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0
catheter site pain (General disorders) | 1 | 0 | 2
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0
Vessel puncture site reaction (General disorders) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Heart Rate increased (Investigations) | 0 | 1 | 1
Mean cell volume increased (Investigations) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hot Flush (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days